CLINICAL TRIAL: NCT06407700
Title: Comparative Effects of Brugger's Exercise With and Without Kendall Exercises on Pain, Craniovertebral Angle and Range of Motion in Patients With Sterno-Symphyseal Syndrome
Brief Title: Comparison of Brugger's Exercise With and Without Kendall Exercises in Sterno-Symphyseal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0185
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Upper Crossed Syndrome
Keywords: Craniovertebral Anglle.; Exercise; Pain; Posture; Sterno-symphyseal Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the treatment arms at the beginning of the trial and continue in that arm throughout the length of the trial.
Who Masked: Outcomes Assessor
Masking Description: Blinding,refers to a practice where study participants are prevented from knowing certain information that may somehow influence them-thereby tainting the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brugger's exercise with Kendall exercise. (Experimental): Participants in this group will receive Brugger's exercise with Kendall Exercise.
  Interventions: Procedure: Brugger's exercise.; Procedure: Kendall Exercise.
- Brugger's exercise (Active Comparator): Participants in this group will receive Brugger's exercise.
  Interventions: Procedure: Brugger's exercise.

INTERVENTIONS:
Procedure: Brugger's exercise. — Participant was in a high sitting position. An elastic resistance band was be wrapped on each hand of the participant leaving the palm open and instructed to abduct and extend of thumb along with fingers, followed by wrist extension and forearm supination, the participant were instructed to perform scapular retraction with chin tucked in ,shoulder external rotation, elbow extension, shoulder abduction, and extension. Intervention was started from 10 seconds hold to 30 seconds with 2 seconds increment in every session. Rest time was 30 seconds, 4 sets 12 times repetitions.
Procedure: Kendall Exercise. — Kendall exercises with the frequency 5 sets of consisting of 12 repetitions of postures, each taking 30 seconds,3 times a week for total of 6 weeks.
  Arms: Brugger's exercise with Kendall exercise.

SUMMARY:
Sterno-symphyseal syndrome is a natural result of prolonged sitting work, especially with computers .In actual it is the approximation between pubic symphysis and sternum. The aim of study will be to compare the effects of Brugger's exercise with and without Kendall exercises on Pain, Craniovertebral angle and Range of motion in patients with Sterno-Symphyseal Syndrome. Group A will be treated with Kendall exercises and Brugger's Exercise and Group B will receive Brugger's Exercise only. Standard treatment will be provided to both groups. Outcome measures will be conducted at baseline, after 3 weeks and by the end of 6 weeks of treatment. Data will be analyzed using SPSS software version 25.

DETAILED DESCRIPTION:
Sterno-symphyseal syndrome is a natural result of prolonged sitting work, especially with computers. It is basically the approximation between the sternum and pubic symphysis. This syndrome has been given several names including posterior cervical-dorsal syndrome and more commonly Computer back or Student syndrome. This posture is associated with increased muscular tension and faulty respiration habit. The aim of study will be to compare the effects of Brugger's exercise with and without Kendall exercises on Pain, Craniovertebral angle and Range of motion in patients with Sterno-Symphyseal Syndrome.

A Randomized Clinical Trial will be conducted at Umar Hospital Lahore through convenience sampling technique on patients which will be allocated using simple random sampling through computer generated method into Group A and Group B. Group A will be treated with Kendall exercises and Brugger's Exercise and Group B will receive Brugger's Exercise only. Standard treatment will be provided to both groups. Outcome measures will be conducted through pain, Craniovertebral angle and neck range of motion at baseline, after 3 weeks and by the end of 6 weeks of treatment. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria: • Age Group between 18-35 years old

* Gender: Male and Female both included (23).
* Subjects with slumped posture with Craniovertebral angle less than 50 degree (12).
* Subjects having distance from xiphoid process to pubic symphysis less than 28 cm (11 inches).
* Subjects sitting more than 4 hours a day (12).
* Subjects with upper back pain with < 7 score on Numeric Pain rating scale

Exclusion Criteria: • Subjects with Untreated fractures on cervical and upper thorax spine.

* Neoplasm on spine.
* Cervical disc prolapses.
* Subject with psychological disorder.
* Vertebro basilar insufficiency and Migraine are excluded (12).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-04 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 6th week.
  Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain". Reliability is 0.76-0.96 .
Measuring tape for Sterno-symphyseal syndrome. | 6th week.
  To measure distance between xiphoid process and pubic symphysis.
Universal Goniometer (UG) | 6th week
  3. Universal Goniometer (UG) It is commonly a large universal goniometer having 12-inch arms and full-circle plastic body used for measuring AROM. It is used to measure joint ROM in clinics. Reliability is 0.9.
  It will measure range of motion of neck. It will measure Craniovertebral angle.
Image J Software | 6th week.
  Image J is an image Processing tool that processes photographs taken for the observation of Posture. Image J, a versatile software, has many capabilities and functions. This software is very simple and easily available. By Using JAVA, it is built on open architecture platform. Validity is 0.96 (31)

CONTACTS AND LOCATIONS:
Overall Officials: Tooba Jamil, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- Umar Trust Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park JH, Moon JH, Kim HJ, Kong MH, Oh YH. Sedentary Lifestyle: Overview of Updated Evidence of Potential Health Risks. Korean J Fam Med. 2020 Nov;41(6):365-373. doi: 10.4082/kjfm.20.0165. Epub 2020 Nov 19. PMID 33242381
- [Background] Damen I, Brombacher H, Lallemand C, Brankaert R, Brombacher A, van Wesemael P, Vos S. A Scoping Review of Digital Tools to Reduce Sedentary Behavior or Increase Physical Activity in Knowledge Workers. Int J Environ Res Public Health. 2020 Jan 13;17(2):499. doi: 10.3390/ijerph17020499. PMID 31941096
- [Background] Romero-Blanco C, Rodriguez-Almagro J, Onieva-Zafra MD, Parra-Fernandez ML, Prado-Laguna MDC, Hernandez-Martinez A. Physical Activity and Sedentary Lifestyle in University Students: Changes during Confinement Due to the COVID-19 Pandemic. Int J Environ Res Public Health. 2020 Sep 9;17(18):6567. doi: 10.3390/ijerph17186567. PMID 32916972
- [Background] Moreira S, Criado MB, Santos PC, Ferreira MS, Goncalves C, Machado J. Occupational Health: Physical Activity, Musculoskeletal Symptoms and Quality of Life in Computer Workers: A Narrative Review. Healthcare (Basel). 2022 Dec 5;10(12):2457. doi: 10.3390/healthcare10122457. PMID 36553981
- [Background] Lee S, DE Barros FC, DE Castro CSM, DE Oliveira Sato T. Effect of an ergonomic intervention involving workstation adjustments on musculoskeletal pain in office workers-a randomized controlled clinical trial. Ind Health. 2021 Mar 24;59(2):78-85. doi: 10.2486/indhealth.2020-0188. Epub 2020 Nov 28. PMID 33250456
- [Background] He M, Wang X, Zhao Y. A calibrated deep learning ensemble for abnormality detection in musculoskeletal radiographs. Sci Rep. 2021 Apr 27;11(1):9097. doi: 10.1038/s41598-021-88578-w. PMID 33907257
- [Background] Waongenngarm P, van der Beek AJ, Akkarakittichoke N, Janwantanakul P. Perceived musculoskeletal discomfort and its association with postural shifts during 4-h prolonged sitting in office workers. Appl Ergon. 2020 Nov;89:103225. doi: 10.1016/j.apergo.2020.103225. Epub 2020 Aug 2. PMID 32755740
- [Background] Gallego-Izquierdo T, Arroba-Diaz E, Garcia-Ascoz G, Val-Cano MDA, Pecos-Martin D, Cano-de-la-Cuerda R. Psychometric Proprieties of a Mobile Application to Measure the Craniovertebral Angle a Validation and Reliability Study. Int J Environ Res Public Health. 2020 Sep 8;17(18):6521. doi: 10.3390/ijerph17186521. PMID 32911612
- [Background] Jung KS, Jung JH, In TS, Cho HY. Effects of Prolonged Sitting with Slumped Posture on Trunk Muscular Fatigue in Adolescents with and without Chronic Lower Back Pain. Medicina (Kaunas). 2020 Dec 23;57(1):3. doi: 10.3390/medicina57010003. PMID 33374520
- [Background] Yoo WG. Effects of thoracic posture correction exercises on scapular position. J Phys Ther Sci. 2018 Mar;30(3):411-412. doi: 10.1589/jpts.30.411. Epub 2018 Mar 2. PMID 29581661
- [Background] Celik S, Celik K, Dirimese E, Tasdemir N, Arik T, Buyukkara I. Determination of pain in musculoskeletal system reported by office workers and the pain risk factors. Int J Occup Med Environ Health. 2018 Jan 1;31(1):91-111. doi: 10.13075/ijomeh.1896.00901. Epub 2017 Oct 2. PMID 28972599
- [Background] Cote R, Vietas C, Kolakowski M, Lombardo K, Prete J, Dashottar A. Inter and Intra-Rater Reliability of Measuring Photometric Craniovertebral Angle Using a Cloud-Based Video Communication Platform. Int J Telerehabil. 2021 Jun 22;13(1):e6346. doi: 10.5195/ijt.2021.6346. eCollection 2021. PMID 34345337
- [Background] Sukari AAA, Singh S, Bohari MH, Idris Z, Ghani ARI, Abdullah JM. Examining the Range of Motion of the Cervical Spine: Utilising Different Bedside Instruments. Malays J Med Sci. 2021 Apr;28(2):100-105. doi: 10.21315/mjms2021.28.2.9. Epub 2021 Apr 21. PMID 33958964
- [Background] Denton F, Power S, Waddell A, Birkett S, Duncan M, Harwood A, McGregor G, Rowley N, Broom D. Is It Really Home-Based? A Commentary on the Necessity for Accurate Definitions across Exercise and Physical Activity Programmes. Int J Environ Res Public Health. 2021 Sep 1;18(17):9244. doi: 10.3390/ijerph18179244. PMID 34501833
- [Background] Yaghoubitajani Z, Gheitasi M, Bayattork M, Andersen LL. Corrective exercises administered online vs at the workplace for pain and function in the office workers with upper crossed syndrome: randomized controlled trial. Int Arch Occup Environ Health. 2022 Oct;95(8):1703-1718. doi: 10.1007/s00420-022-01859-3. Epub 2022 Apr 7. PMID 35391580
- [Background] Mylonas K, Angelopoulos P, Billis E, Tsepis E, Fousekis K. Combining targeted instrument-assisted soft tissue mobilization applications and neuromuscular exercises can correct forward head posture and improve the functionality of patients with mechanical neck pain: a randomized control study. BMC Musculoskelet Disord. 2021 Feb 21;22(1):212. doi: 10.1186/s12891-021-04080-4. PMID 33612123
- [Background] Chang KV, Wu WT, Chen MC, Chiu YC, Han DS, Chen CC. Smartphone Application with Virtual Reality Goggles for the Reliable and Valid Measurement of Active Craniocervical Range of Motion. Diagnostics (Basel). 2019 Jul 10;9(3):71. doi: 10.3390/diagnostics9030071. PMID 31295869